CLINICAL TRIAL: NCT02780128
Title: Next Generation Personalized Neuroblastoma Therapy (The NEPENTHE Trial)
Brief Title: Next Generation Personalized Neuroblastoma Therapy
Acronym: NEPENTHE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The goals of Part 1 (molecular screening) were met, but lack of therapies to match molecular aberrations made Part 2 (treatment) no longer feasible.
Sponsor: Yael P Mosse (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Foundation Medicine (Industry)
Responsible Party: Sponsor-Investigator, Yael P Mosse, Principal Investigator, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-011071
Record Dates: First submitted 2016-05-11; First posted 2016-05-23 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Neuroblastoma; Cancer
Keywords: neuroblastoma; cancer; genetic profiling; ceritinib; ribociclib; NEPENTHE
MeSH Terms: conditions — Neuroblastoma; Neoplasms | interventions — Biopsy; High-Throughput Nucleotide Sequencing; Restraint, Physical; Hematologic Tests; Pregnancy Tests; Interviews as Topic; ribociclib; ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Molecular Analysis (Other): All participants with relapsed or refractory neuroblastoma will have a tumor biopsy to identify genetic mutations. There is no drug given in this arm of the trial.
  Interventions: Procedure: Biopsy; Genetic: Next Generation Sequencing; Procedure: Tumor Scans; Other: Physical Exam; Other: Labs; Other: Pregnancy Test; Behavioral: Interviews
- Group 1: ALK (Experimental): Qualified participants whose tumors show certain mutations in the anaplastic lymphoma kinase (ALK) pathway (based on genetic sequencing results) will receive a combination therapy of ceritinib and ribociclib, to be administered orally in 28-day cycles.
  Two different doses of ceritinib and three different doses of ribociclib will be evaluated. Once the investigators have identified the highest safe dose of both drugs that can be given at the same time, additional participants will be enrolled in the study at this dose level.
  It is possible that if starting at a lower dose, participants may take a higher dose once that dose has been deemed safe.
  Interventions: Procedure: Tumor Scans; Procedure: Bone marrow Tests; Other: Physical Exam; Other: Eye Exam; Other: Labs; Other: Pregnancy Test; Behavioral: Interviews; Other: ECG; Other: Echocardiogram; Drug: Ribociclib; Drug: Ceritinib

INTERVENTIONS:
Procedure: Biopsy — Needle or incisional tumor biopsy
  Other Names: Genetic Sequencing
  Arms: Molecular Analysis
Genetic: Next Generation Sequencing — Tumor tissue will be sent to Foundation Medicine laboratory for molecular profiling.
  Other Names: Molecular Profiling; Genetic Sequencing
  Arms: Molecular Analysis
Procedure: Tumor Scans — Participants will undergo different types of scans to look at your tumor. These scans include CT (computerized tomography), MIBG (meta-iodobenzylguanidine) PET (positron emission tomography), and MRI (magnetic resonance imaging). Participants may have more than one type of scan.
Procedure: Bone marrow Tests — Participants will have needles inserted through their hip bone to remove fluid from inside the bone marrow. This test determines if participants have tumor in the bone marrow.
  Other Names: Bone marrow aspiration
  Arms: Group 1: ALK
Other: Physical Exam — The exam includes taking participant weight, height, blood pressure, heart rate and respiratory rate and performing a examination of the participants body. The investigators may also check the participants vision with an eye chart.
Other: Eye Exam — Participants will have their eyes will be evaluated using different instruments. Participants will also be asked to read an eye chart. The exams will take about 15 minutes.
  Other Names: Ophthalmic Exam
  Arms: Group 1: ALK
Other: Labs — Standard blood tests will be done to measure different types of blood cells, to measure the amount of certain substances, and tests to check how well liver and kidneys are working. When possible, the investigators will take blood from the participants central line. If this is not possible, the investigators will take blood from a vein in the participants arm. First, the investigators will put some cream on the skin so that drawing blood will not be painful. Then the investigators will put a thin needle into the vein to draw the blood.
  Other Names: Blood tests
Other: Pregnancy Test — If the participant is 11 years old or older or has already started having periods, the participant will be asked to take a pregnancy test before starting this study. The results will be shared with the participant but not with the participants' parent(s). We strongly encourage the participant to share the results with the parents. If the participant is found to be pregnant, the participant will not be able to continue participation in the study. About 1 teaspoon of blood (or urine if a urine test) will be needed.
Behavioral: Interviews — A team member will take the participant's medical history, along with a listing of any medications that are being taken. Throughout the study, participants will be asked to report if they think that anything bad has happened as a result of the study.
Other: ECG — This is a test of electrical activity of the heart. The investigators will put electrodes (sticky pads attached to wires) on the participant's chest, arms and legs. The electrocardiogram (ECG) will not be uncomfortable, but the participant will have to lie still. It does not hurt and takes about 15 minutes.
  Other Names: EKG; Electrocardiogram
  Arms: Group 1: ALK
Other: Echocardiogram — The participant will have an Echocardiogram (ECHO), an ultrasound of the heart, taken to assess heart function. The investigators will put some gel on the skin and use a machine to take pictures of the heart.
  Other Names: ECHO
  Arms: Group 1: ALK
Drug: Ribociclib — Participants will take ribociclib once per day orally for Days 1-21 of a 28-day cycle.
  Other Names: LEE011
  Arms: Group 1: ALK
Drug: Ceritinib — Participants will take ceritinib once per day orally for 28 days of a 28-day cycle.
  Other Names: LDK378
  Arms: Group 1: ALK

SUMMARY:
The purpose of this research study is to match genomic aberrations in tumor cells at time of relapse to rationally designed combinations of molecularly targeted agents. This study will be done in two parts:

Part I: Tumor will be accessed at study entry via a biopsy and subjected to deep sequencing to identify protocol-specified biomarkers for therapy assignment.

Part II: If the tumor contains a genetic change defined by the study as being actionable, and other criteria are met, participants will be assigned to therapy based upon the genetic changes identified in the tumor biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥1 years to ≤ 21 years
* Relapsed or refractory neuroblastoma
* A sufficient interval between the last dose of prior anti-cancer therapy (including cytotoxic and biological therapies) and enrollment in this study, to allow recovery from the acute toxic effects of all prior anti-cancer therapy. Please contact site for specific details
* Adequate bone marrow function (bone marrow may be involved with tumor. Contact site for specific details)
* Adequate renal function, defined as Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 70 mL/min/1.73 m2 OR serum creatinine based on age/gender normal (contact site for details)
* Adequate liver function, defined as total serum bilirubin ≤ 1.5 times the upper limit of normal AND alanine transaminase (ALT) ≤ 110 U/L.
* Adequate cardiac function, defined as corrected QT interval (QTc) ≤ 480 msec AND shortening fraction > 27%
* Males and females who are sexually active must agree to use effective contraception during and for 3 months after treatment

Exclusion Criteria:

* Subjects taking certain drugs or herbal medications that impact drug metabolism and/or cardiac function that cannot be discontinued (contact site for details).
* Subjects with concurrent severe and/or uncontrolled concurrent medical conditions that could compromise participation in the study (contact site for details)
* Other concomitant therapies:
* Corticosteroids initiated for tumor therapy within 7 days prior to study enrollment
* Other anti-cancer agents
* Other investigational drugs
* Hematological growth factors
* Radiation therapy
* Subjects < 0.5m2
* Pregnant or lactating females
* Sexually active males unless they use a condom during intercourse while taking study drug/s and for 3 months after study drug discontinuation and thus do not attempt to father a child in this period.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities when combining ceritinib with ribociclib | At the end of Cycle 1 (each cycle is 28 days)
  The primary variable is the incidence of dose limiting toxicities (DLTs) during the first 28 days of therapy
Area under the curve from time zero to last quantifiable concentration | At the end of Cycle 1 (each cycle is 28 days)
  Area under the plasma concentration time-curve from zero to the last measured concentration
Percentage of patients with overall objective response | 2 years
  To describe whether the assigned targeted therapy can mediate anti-tumor effects in subjects with relapsed or refractory high-risk neuroblastoma within the context of a phase 1/phase1b biomarker-driven trial. Percentage of patients with objective response will be according to the International Neuroblastoma Response Criteria.

SECONDARY OUTCOMES:
Cataloguing of genomic alterations identified from biopsies performed at time of relapse in patients with relapsed or refractory neuroblastoma | 3 years
  Neuroblastomas undergo substantial mutational evolution during therapy, and relapsed disease is more likely to be driven by a targetable oncogenic pathway. Genomic alterations measured by next-generation sequencing at time of disease progression will be characterized and reported in a descriptive manner.

CONTACTS AND LOCATIONS:
Overall Officials: Yael P Mossé, MD, Principal Investigator — Children's Hospital of Philadelphia, The University of Pennsylvania; John M Maris, MD, Principal Investigator — Children's Hospital of Philadelphia, The University of Pennsylvania
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Rader J, Russell MR, Hart LS, Nakazawa MS, Belcastro LT, Martinez D, Li Y, Carpenter EL, Attiyeh EF, Diskin SJ, Kim S, Parasuraman S, Caponigro G, Schnepp RW, Wood AC, Pawel B, Cole KA, Maris JM. Dual CDK4/CDK6 inhibition induces cell-cycle arrest and senescence in neuroblastoma. Clin Cancer Res. 2013 Nov 15;19(22):6173-82. doi: 10.1158/1078-0432.CCR-13-1675. Epub 2013 Sep 17. PMID 24045179
- [Background] Bresler SC, Weiser DA, Huwe PJ, Park JH, Krytska K, Ryles H, Laudenslager M, Rappaport EF, Wood AC, McGrady PW, Hogarty MD, London WB, Radhakrishnan R, Lemmon MA, Mosse YP. ALK mutations confer differential oncogenic activation and sensitivity to ALK inhibition therapy in neuroblastoma. Cancer Cell. 2014 Nov 10;26(5):682-94. doi: 10.1016/j.ccell.2014.09.019. Epub 2014 Nov 10. PMID 25517749
- [Background] Bresler SC, Wood AC, Haglund EA, Courtright J, Belcastro LT, Plegaria JS, Cole K, Toporovskaya Y, Zhao H, Carpenter EL, Christensen JG, Maris JM, Lemmon MA, Mosse YP. Differential inhibitor sensitivity of anaplastic lymphoma kinase variants found in neuroblastoma. Sci Transl Med. 2011 Nov 9;3(108):108ra114. doi: 10.1126/scitranslmed.3002950. PMID 22072639
- [Background] Carr-Wilkinson J, O'Toole K, Wood KM, Challen CC, Baker AG, Board JR, Evans L, Cole M, Cheung NK, Boos J, Kohler G, Leuschner I, Pearson AD, Lunec J, Tweddle DA. High Frequency of p53/MDM2/p14ARF Pathway Abnormalities in Relapsed Neuroblastoma. Clin Cancer Res. 2010 Feb 15;16(4):1108-18. doi: 10.1158/1078-0432.CCR-09-1865. Epub 2010 Feb 9. PMID 20145180
- [Background] Geoerger B, Bourdeaut F, DuBois SG, Fischer M, Geller JI, Gottardo NG, Marabelle A, Pearson ADJ, Modak S, Cash T, Robinson GW, Motta M, Matano A, Bhansali SG, Dobson JR, Parasuraman S, Chi SN. A Phase I Study of the CDK4/6 Inhibitor Ribociclib (LEE011) in Pediatric Patients with Malignant Rhabdoid Tumors, Neuroblastoma, and Other Solid Tumors. Clin Cancer Res. 2017 May 15;23(10):2433-2441. doi: 10.1158/1078-0432.CCR-16-2898. Epub 2017 Apr 21. PMID 28432176
- [Background] Hart LS, Rader J, Raman P, Batra V, Russell MR, Tsang M, Gagliardi M, Chen L, Martinez D, Li Y, Wood A, Kim S, Parasuraman S, Delach S, Cole KA, Krupa S, Boehm M, Peters M, Caponigro G, Maris JM. Preclinical Therapeutic Synergy of MEK1/2 and CDK4/6 Inhibition in Neuroblastoma. Clin Cancer Res. 2017 Apr 1;23(7):1785-1796. doi: 10.1158/1078-0432.CCR-16-1131. Epub 2016 Oct 11. PMID 27729458
- [Background] Mosse YP, Laudenslager M, Longo L, Cole KA, Wood A, Attiyeh EF, Laquaglia MJ, Sennett R, Lynch JE, Perri P, Laureys G, Speleman F, Kim C, Hou C, Hakonarson H, Torkamani A, Schork NJ, Brodeur GM, Tonini GP, Rappaport E, Devoto M, Maris JM. Identification of ALK as a major familial neuroblastoma predisposition gene. Nature. 2008 Oct 16;455(7215):930-5. doi: 10.1038/nature07261. Epub 2008 Aug 24. PMID 18724359
- [Background] Mosse YP, Lim MS, Voss SD, Wilner K, Ruffner K, Laliberte J, Rolland D, Balis FM, Maris JM, Weigel BJ, Ingle AM, Ahern C, Adamson PC, Blaney SM. Safety and activity of crizotinib for paediatric patients with refractory solid tumours or anaplastic large-cell lymphoma: a Children's Oncology Group phase 1 consortium study. Lancet Oncol. 2013 May;14(6):472-80. doi: 10.1016/S1470-2045(13)70095-0. Epub 2013 Apr 16. PMID 23598171
- [Background] Mosse YP, Voss SD, Lim MS, Rolland D, Minard CG, Fox E, Adamson P, Wilner K, Blaney SM, Weigel BJ. Targeting ALK With Crizotinib in Pediatric Anaplastic Large Cell Lymphoma and Inflammatory Myofibroblastic Tumor: A Children's Oncology Group Study. J Clin Oncol. 2017 Oct 1;35(28):3215-3221. doi: 10.1200/JCO.2017.73.4830. Epub 2017 Aug 8. PMID 28787259
- [Background] Padovan-Merhar OM, Raman P, Ostrovnaya I, Kalletla K, Rubnitz KR, Sanford EM, Ali SM, Miller VA, Mosse YP, Granger MP, Weiss B, Maris JM, Modak S. Enrichment of Targetable Mutations in the Relapsed Neuroblastoma Genome. PLoS Genet. 2016 Dec 20;12(12):e1006501. doi: 10.1371/journal.pgen.1006501. eCollection 2016 Dec. PMID 27997549
- [Background] Rihani A, Vandesompele J, Speleman F, Van Maerken T. Inhibition of CDK4/6 as a novel therapeutic option for neuroblastoma. Cancer Cell Int. 2015 Jul 30;15:76. doi: 10.1186/s12935-015-0224-y. eCollection 2015. PMID 26225123
- [Background] Van Maerken T, Rihani A, Dreidax D, De Clercq S, Yigit N, Marine JC, Westermann F, De Paepe A, Vandesompele J, Speleman F. Functional analysis of the p53 pathway in neuroblastoma cells using the small-molecule MDM2 antagonist nutlin-3. Mol Cancer Ther. 2011 Jun;10(6):983-93. doi: 10.1158/1535-7163.MCT-10-1090. Epub 2011 Apr 1. PMID 21460101
- [Background] Van Maerken T, Vandesompele J, Rihani A, De Paepe A, Speleman F. Escape from p53-mediated tumor surveillance in neuroblastoma: switching off the p14(ARF)-MDM2-p53 axis. Cell Death Differ. 2009 Dec;16(12):1563-72. doi: 10.1038/cdd.2009.138. Epub 2009 Sep 25. PMID 19779493
- [Background] Wood AC, Krytska K, Ryles HT, Infarinato NR, Sano R, Hansel TD, Hart LS, King FJ, Smith TR, Ainscow E, Grandinetti KB, Tuntland T, Kim S, Caponigro G, He YQ, Krupa S, Li N, Harris JL, Mosse YP. Dual ALK and CDK4/6 Inhibition Demonstrates Synergy against Neuroblastoma. Clin Cancer Res. 2017 Jun 1;23(11):2856-2868. doi: 10.1158/1078-0432.CCR-16-1114. Epub 2016 Dec 16. PMID 27986745